CLINICAL TRIAL: NCT05243784
Title: The Impact of a Classroom-based Physical Activity Breaks on Cognitive Function, Adiposity and Fitness in Preschool Children. A Pilot Trial Study (MOVI- HIIT)
Brief Title: The MOVI-HIIT Pilot Trial: The Impact of Activity Breaks on Cognitive Function, Adiposity and Fitness in Preschoolers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Castilla-La Mancha (Other)
Collaborators: Ministerio de Ciencia e Innovación, Spain (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: PID2019-104160RB-I00-Pilot
Record Dates: First submitted 2022-01-03; First posted 2022-02-17 (Actual); Last update posted 2022-11-03 (Actual); Status verified 2022-11

CONDITIONS: Physical Activity; Obesity, Childhood; Cardiovascular Diseases; High Intensity Interval Training; Cognition
Keywords: Children; obesity; High Intensity Interval Training; cognition; cardiorespiratory fitness; Aerobic capacity; Preschool; Adiposity; Physical Activity
MeSH Terms: conditions — Motor Activity; Pediatric Obesity; Cardiovascular Diseases; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): The design of the MOVI-HIIT intervention is framed within the socio-ecological model of behavior modification, in such a way that it will be designed to intervene in the individual, family and school environment. It will have a duration of 8 weeks and will consist of two 5-minute daily physical activity breaks based on intervallic training, five days a week.
  Interventions: Behavioral: MOVI-HIIT intervention
- Control (No Intervention): Students in the control group (CG) will receive mandatory lessons on Spain (one 45-minute session of Psychomotor/Physical Education), and the usual classroom teaching methodology. Teachers in the CG schools will be asked not to make any changes to their methodology during the time of the study, with the promise by the research team to share and explain the MOVI-HIIT program once the interventions are completed.

INTERVENTIONS:
Behavioral: MOVI-HIIT intervention — Each HIIT break will last approximately 5 minutes and will not require any specific materials. The structure of the HIIT-Rest will be as follows: 1' to describe the work to be done; 3' of work following the HIIT protocol: 6 repetitions of a functional movement such as squats, Jumping Jack or running on site for 20" at high intensity (85-90% of HR -heart rate- max) followed by 10" of recovery (65-75% of HR max); and 1' to perform a return to calm in order to lower the activation and prepare the student body to return to class activities.
  Arms: Intervention

SUMMARY:
Pilot study to test the acceptability and feasibility of an intervention aimed to test the effectiveness, in preschool children, of an integrated physical activity intervention in the classroom based on intervallic training (MOVI-HIIT) on improving executive function, body composition and cardiorespiratory fitness.

DETAILED DESCRIPTION:
The evolution of the MOVI studies, conducted by the research group, has led to create the last project (MOVI-HIIT; ClinicalTrials.gov Identifier: NCT04863040).

This pilot study will include children aged 4-6 years from 2 public schools of the province of Ciudad Real, Spain, with 2 arms (intervention and control) and the intervention will last 8 weeks.

The intervention proposed in the study is implemented through an online platform developed to achieved the intensities required for the age-range of participants, but this platform has never been tested accurately in the classroom.

Thus, it seems necessary to pilot the intervention to evaluate the acceptability and feasibility of the intervention, in order to improve facts, if necessary, to achieved proposed objectives.

ELIGIBILITY:
Inclusion Criteria:

* The participating schoolchildren must belong to the 2nd and 3rd year of preschool education, not have any malformation that prevents them from learning the Spanish language (or Spanish sign language), not have any type of physical or mental disorder that parents and/or teachers have identified that prevents the performance of physical activities, not suffer from any chronic disease such as heart disease, diabetes or asthma that, according to the criteria of their pediatrician - after analysis of the program of activities - prevents their participation in the measurements and/or the intervention.
* As this is an intervention in the classroom, the school faculty will include the active breaks proposed in the center's programming, for which reason the intervention will be received by all the children in the intervention group school. However, the investigators will consider school participants to be those who have the consent of the parent or guardian for participation in the study. In addition, schoolchildren must verbally express their willingness to participate in the baseline and final physical examinations.

Exclusion Criteria:

* Children with severe Spanish language learning difficulties.
* Children with serious physical or mental disorders identified by parents or teachers that would impede participation in the programme's activities.
* Children diagnoses of chronic disorders, such as heart disease, diabetes or asthma, which in the opinion of their paediatricians would prevent their participation in the programme's activities (MOVI-HIIT)

Ages: 4 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 62 (Actual)
Dates: Start 2022-01-27 (Actual); Primary Completion 2022-04-01 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Evaluation of the perceived effort and exercise enjoyment within the use of the MOVI-HIIT platform by questionnaires. | 4 months
  The schoolchildren's exercise enjoyment will be measured with the short version of the Physical Activity Enjoyment Scale, PACES-S [10.3390/ijerph182111035]), (range from 4 to 12, where the highest rate indicates more satisfaction); and the schoolchildren's perceived effort will be assessed with the Children's Effort Rating Table, Pictorial-CERT [10.1111/j.1365-2214.2007.00767.x.], with a range from 1 to 10 (where 10 indicates the highest perceived effort).
Acceptance rate and adverse effects of the MOVI-HIIT intervention. | 4 months
  The acceptability of the exercise program will be assessed recording adherence (rate of school's session attendance recorded in the online platform) and safety of the exercise programme (number and type of adverse events recorded by the teacher everyday after the session).
Evaluation of schoolchildren's compliance with the MOVI-HIIT intervention. | 4 months
  These trial feasibility outcomes will include: (1) recruitment (percentage achieved of the targeted study sample), (2) retention (drop-out rate and reasons for withdrawal), (3) outcome completion (percentage of children with both measurements at the end of the study).
Participant's satisfaction with the MOVI-HIIT program by questionnaire | 4 months
  An ad-hoc questionnarie will ask participants' about their satisfaction with the program (5-item pictorial scale questions, where the higher rate indicates higher satisfaction).
Teacher's perception about the suitability of the MOVI-HIIT platform by interviews. | 4 months
  It will be assessed with teachers feedback via interviews on the use of the exercise platform (user-friendliness, connectivity, attractiveness, practicality) and the barriers and facilitators to implementing the programme.

SECONDARY OUTCOMES:
VO2max | 4 months
  Cardiorespiratory fitness (Course Navette or 20-m shuttle run test), validated to measure maximum aerobic capacity in children. It will be carried out according to the Léger protocol included in the PREFIT Battery: Assessing FITness in PREschoolers adapted to children under the age of 6.
Inhibition/Attention (Executive Function) | 4 months
  Measured by means of the Flanker Inhibitory Control and Attention test included in the NIH toolbox battery.
Working memory (Executive Function) | 4 months
  Working memory with the Word Span test included in the NIH toolbox battery. This test is the Spanish version of the procedure developed by Thorell and Wählstedt (2006), based on the Digit Span subtest from the Wechsler Intelligence Test for Children-3rd edition (WISC-III; Wechsler, 1991).
Cognitive flexibility (Executive Function) | 4 months
  NIH toolbox battery. Cognitive flexibility through the DCCS (Dimensional Change Card Sort) test, included in the NIH toolbox battery.
Percentage of body fat | 4 months
  It will be measured twice in each participant by bioimpedance analysis.
Health Related Quality of Life for children and parents | 4 months
  Kiddy-KINDL-R questionnaire version for children and parents accordingly, which has a 0-100 score scale (the higher score, the better perceived quality of life).
Amount of daily performed physical activity | 4 months
  Physical activity will be objectively measured with pedometers during the day at school and in three moments across the pilot project (before, during and after the intervention).
The acute effect of physical exercise on the brain's electrical activity | 4 months
  The brain activity will be measured with a portable electroencephalogram (EMOTIV EPOC X - 14-channel EEG - for whole brain sensing (AF3, AF4, F3, F4, F7, F8, T7, T8, P3, P4, P7, P8, O1, O2)) in 30 schoolchildren (15 children in the intervention group and 15 in the control group).
Children's active commuting to school questionnaire | 4 months
  Patterns of commuting to school will be collected through a questionnaire for the children's parents, including 2 questions about the mode and duration of the commute to school: (1) ''How does your son/daughter usually go from home to school?'' and (2) ''How long does it usually take for your son/daughter to go from home to school?''. These questions are obtained from a 7-item questionnaire whose validity and reliability have been shown (Evenson KR et al. J Phys Act Health. 2008;5(suppl 1):S1-S15).

CONTACTS AND LOCATIONS:
Locations (1):
- Social and Health Research Center. Universidad de Castilla-La Mancha, Cuenca, Spain

IPD SHARING:
Plan to Share IPD: No